CLINICAL TRIAL: NCT03071237
Title: The Origin of Infrapyloric Artery: an Observational Trial
Brief Title: The Origin of Infrapyloric Artery
Acronym: IPA-Origin
Status: Completed | Type: Observational
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, Jiafu Ji, MD, Peking University
Other Study IDs: 2017YJZ07
Record Dates: First submitted 2017-03-01; First posted 2017-03-06 (Actual); Last update posted 2019-02-19 (Actual); Status verified 2019-02

CONDITIONS: Stomach Neoplasm
Keywords: infrapyloric artery; gastric cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — Gastrectomy; Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational group: Patients who would receive total gastrectomy or distal gastrectomy are enrolled in to the study and this group. An optional reconstruction of IPA by enhanced CT scan can be performed before surgery but not a definite require. During the operation, IPA origin location will be photo-taken or video-recorded before its transection.
  Interventions: Procedure: Gastrectomy

INTERVENTIONS:
Procedure: Gastrectomy — Patients with gastric cancer that needs receiving total or distal gastrectomy. During the surgery, IPA needs to be exposed and transected.
  Other Names: surgery

SUMMARY:
Infrapyloric artery(IPA) is of great importance for gastric cancer patients. According to previous study, the origin of IPA varies greatly among different studies. This trial aims to tell the distribution of IPA origin in Chinese patients.

DETAILED DESCRIPTION:
Infrapyloric artery(IPA) is of great importance for gastric cancer patients. In early gastric cancer patients, the pylorus-preserving gastrectomy requires the preserving of IPA. In advanced gastric cancer patients, the subgroup of No. 6 lymph node might be associated with IPA. In Japanese Gastric Cancer Association(JGCA) gastric cancer classification guidelines, the No. 6 lymph nodes is defined as lymph nodes along the first branch and proximal part of the right gastroepiploic artery(RGEA) down to the confluence of the right gastroepiploic vein and the anterior superior pancreatoduodenal vein. However,if IPA origins from the gastroduodenal artery(GDA) or anterior superior pancreatoduodenal artery(ASPDA), the lymph nodes along the IPA can not be grouped into the No. 6 lymph nodes. Thus, a new definition of No. 6 lymph nodes is needed on the basis of the origin of IPA.

Previous studies about IPA origin are few and the origin of IPA varies greatly among different studies.

ELIGIBILITY:
Inclusion Criteria:

* Patients with gastric cancer who needs to receive total or distal gastrectomy.
* Signed informed consent

Exclusion Criteria:

* IPA not dissected, photo-taken or video-recorded.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with gastric cancer who needs to receive total or distal gastrectomy.
Sampling Method: Probability Sample
Enrollment: 429 (Actual)
Dates: Start 2017-03-04 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Distribution of IPA origin | Immediately after surgery
  The percentage of IPA origin from GDA, ASPDA and RGEA.

SECONDARY OUTCOMES:
Reconstruction rate of IPA by CT scan | Immediately after the reconstruction of CT scan.
  The rate of identification of IPA origin by reconstruction of CT scan.

CONTACTS AND LOCATIONS:
Overall Officials: Ziyu Li, M.D., Principal Investigator — Gastrointestinal Cancer Center, Peking University
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Haruta S, Shinohara H, Ueno M, Udagawa H, Sakai Y, Uyama I. Anatomical considerations of the infrapyloric artery and its associated lymph nodes during laparoscopic gastric cancer surgery. Gastric Cancer. 2015 Oct;18(4):876-80. doi: 10.1007/s10120-014-0424-5. Epub 2014 Sep 17. PMID 25228163
- [Background] Shinohara H, Kurahashi Y, Kanaya S, Haruta S, Ueno M, Udagawa H, Sakai Y. Topographic anatomy and laparoscopic technique for dissection of no. 6 infrapyloric lymph nodes in gastric cancer surgery. Gastric Cancer. 2013 Oct;16(4):615-20. doi: 10.1007/s10120-012-0229-3. Epub 2013 Jan 13. PMID 23314832
- [Derived] Miao R, Qu J, Li Z, Wang D, Yu J, Zang W, Li Y, Liu F, Zhang J, Song W, Ye K, Yan S, Wang W, Ren S, Zang L, Jing C, Zhang L, Wang K, Fu W, Fan L, Liang B, Zhao G, Cai J, Yang L, Zhu J, You J, Yang K, Huang Q, Niu Z, Ning N, Qiu X, Ji G, Liang F, Huang H, Gao C, Shan F, Li S, Jia Y, Zhang L, Ying X, Zhang Y, Bu Z, Su X, Zhao G, Li Z, Ji J. Anatomical variation of infra-pyloric artery origination: A prospective multicenter observational study (IPA-Origin). Chin J Cancer Res. 2018 Oct;30(5):500-507. doi: 10.21147/j.issn.1000-9604.2018.05.03. PMID 30510361